CLINICAL TRIAL: NCT04321252
Title: A Randomized, Subject and Investigator-blinded, Placebo Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of KAE609 Administered Intravenously in Healthy Subjects
Brief Title: Study to Assess Safety, Tolerability and Phamacokinetics of KAE609 Administered Intravenously in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CKAE609X2111; 2019-000405-71 (EudraCT Number); 217692/Z/19/Z (Other Grant/Funding Number: Wellcome Trust Grant Number)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-10

CONDITIONS: Malaria
Keywords: safety; tolerability; pharmacokinetics; healthy volunteers; phase 1; malaria; intravenous; iv; KAE609; Placebo
MeSH Terms: conditions — Malaria | interventions — NITD 609

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort A1: 10.5 mg/placebo (Experimental): Single iv bolus dose of KAE609 or placebo administered at the clinical site by the study personnel.
  Interventions: Drug: KAE609; Drug: Placebo
- Cohort A2: 30 mg/placebo (Experimental): Single iv bolus dose of KAE609 or placebo administered at the clinical site by the study personnel.
  Interventions: Drug: KAE609; Drug: Placebo
- Cohort A3: 75 mg/placebo (Experimental): Single iv infusion dose of KAE609 or placebo administered at the clinical site by the study personnel.
  Interventions: Drug: KAE609; Drug: Placebo
- Cohort A4: 120 mg/placebo (Experimental): Single iv infusion dose of KAE609 or placebo administered at the clinical site by the study personnel.
  Interventions: Drug: KAE609; Drug: Placebo
- Cohort A5: 210 mg/placebo (Experimental): Single iv infusion dose of KAE609 or placebo administered at the clinical site by the study personnel.
  Interventions: Drug: KAE609; Drug: Placebo
- Cohort B1: 60 mg/placebo, every 24 hours (q24h) × 5 days (Experimental): Multiple iv bolus doses of KAE609 or placebo administered at the clinical site by the study personnel.
  Interventions: Drug: KAE609; Drug: Placebo
- Cohort B2: 120 mg/placebo, every 24 hours (q24h) × 5 days (Experimental): Multiple iv infusion doses of KAE609 or placebo administered at the clinical site by the study personnel.
  Interventions: Drug: KAE609; Drug: Placebo

INTERVENTIONS:
Drug: KAE609 — * iv bolus administration over approximately 2 min for doses < 75 mg (Cohorts A1, A2 and B1)
  * iv infusion over approximately 10 min for doses ≥ 75 mg (Cohorts A3, A4, A5 and B2)
Drug: Placebo — matching placeo for iv administration

SUMMARY:
This was a randomized, subject and investigator-blinded, placebo-controlled, single and multiple ascending intravenous (iv) dose study in healthy subjects to assess the safety and tolerability of KAE609 given in the vein.

DETAILED DESCRIPTION:
The study consisted of 2 parts: single-ascending dose (SAD) part and multiple ascending dose (MAD) part.

In Part A (Single-ascending dose (SAD) part), it was planned to recruit 6 active, 2 placebo subjects in each cohort:

* Cohort A1: 10.5 mg/placebo
* Cohort A2: 30 mg/placebo
* Cohort A3: 75 mg/placebo
* Cohort A4: 120 mg/placebo
* Cohort A5: 210 mg/placebo

In Part B (Multiple-ascending dose (MAD) part), Subjects were assigned to one of the following treatment arms in a ratio of 2:1 (6 active, 3 placebo):

* Cohort B1: 60 mg/placebo, every 24 hours (q24h) × 5 days
* Cohort B2: 120 mg/placebo, every 24 hours (q24h) × 5 days

Eligible subjects were randomized to receive a single or q24h x 5 doses of either KAE609 or placebo. Safety, tolerability and pharmacokinetics were assessed over the period of 8 days for single dose and 12 days for multiple dose up to end of study visit for each subject.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and female subjects 18 to 55 years of age inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests.
* Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18.0 - 30.0 kg/m2.

Key Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives of Screening, or within 30 days of dosing, whichever is longer; or longer if required by local regulations.
* Significant illness which has not resolved within two (2) weeks prior to initial dosing.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Sexually active males unwilling to use a condom during intercourse while taking investigational drug and for at least 2 weeks after last dose of investigational drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venishetty VK, Lecot J, Nguyen A, Zhang J, Prince WT. First-in-human, randomized, double-blind, placebo-controlled, single and multiple ascending doses clinical study to assess the safety, tolerability, and pharmacokinetics of cipargamin administered intravenously in healthy adults. Antimicrob Agents Chemother. 2024 Sep 4;68(9):e0128723. doi: 10.1128/aac.01287-23. Epub 2024 Jul 26. PMID 39058022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in one center in Belgium.
Groups:
- Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg): Cohort A1 (SAD): Single iv bolus dose of KAE609 10.5 mg administered at the clinical site by the study personnel.
- Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg): Cohort A2 (SAD): Single iv bolus dose of KAE609 30 mg administered at the clinical site by the study personnel.
- Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg): Cohort A3 (SAD): Single iv infusion dose of KAE609 75 mg administered at the clinical site by the study personnel.
- Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg): Cohort A4 (SAD): Single iv infusion dose of KAE609 120 mg administered at the clinical site by the study personnel.
- Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg): Cohort A5 (SAD): Single iv infusion dose of KAE609 210 mg administered at the clinical site by the study personnel.
- Part A (Single-ascending Dose (SAD): Pooled Placebo: All placebo-treated patients from Part A (Single-ascending dose (SAD) cohorts (cohort A1, cohort A2, cohort A3, cohort A4 and cohort A5)
- Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg): Cohort B1 (MAD): Multiple iv bolus doses of KAE609 (60 mg, every 24 hours (q24h) × 5 days) administered at the clinical site by the study personnel.
- Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg): Cohort B2 (MAD): Multiple iv infusion doses of KAE609 (120 mg, every 24 hours (q24h) × 5 days) administered at the clinical site by the study personnel.
- Part B (Multiple-ascending Dose (MAD): Pooled Placebo: All placebo-treated patients from Part B (Multiple-ascending dose (MAD) cohorts (cohort B1 and cohort B2)
Period: Overall Study
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg) | Part A (Single-ascending Dose (SAD): Pooled Placebo | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg) | Part B (Multiple-ascending Dose (MAD): Pooled Placebo
Started (All enrolled participants were included in the Randomized Set and in the Safety Analysis Set) | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
PK Analysis Set (All KAE609-treated participants were included in the PK analysis set) | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg) | Part A (Single-ascending Dose (SAD): Pooled Placebo | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg) | Part B (Multiple-ascending Dose (MAD): Pooled Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 57
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 5 | 16
  Male | 5 | 4 | 5 | 5 | 5 | 7 | 5 | 4 | 1 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 57
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With On-Treatments Adverse Events, Serious Adverse Events, and Deaths
Description: The distribution of adverse events was done via the analysis of frequencies for Adverse Event (AEs), Serious Adverse Event (SAEs) and Deaths, through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From study treatment start date till 30 days safety follow-up, assessed for up to 4 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Part A (Single-ascending Dose (SAD): Pooled KAE609: All KAE609-treated patients from Part A (Single-ascending dose (SAD) cohorts (cohort A1, cohort A2, cohort A3, cohort A4 and cohort A5)
- Part B (Multiple-ascending Dose (MAD): Pooled KAE609: All KAE609-treated patients from Part B (Multiple-ascending dose (MAD) cohorts (cohort B1 and cohort B2)
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg) | Part A (Single-ascending Dose (SAD): Pooled KAE609 | Part A (Single-ascending Dose (SAD): Pooled Placebo | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg) | Part B (Multiple-ascending Dose (MAD): Pooled KAE609 | Part B (Multiple-ascending Dose (MAD): Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30 | 9 | 6 | 6 | 12 | 6
Participants
  Adverse Events (AEs) | 0 | 1 | 1 | 2 | 6 | 10 | 5 | 4 | 6 | 10 | 4
  Serious Adverse Events (SAEs) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Part A - Pharmacokinetic of KAE609: Maximum Observed Plasma Concentration (Cmax)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Cmax was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Day 1 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: PK analysis set. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 412 (101) | 1510 (1000) | 2910 (1340) | 5930 (1190) | 6590 (1290)

3. Secondary Outcome: Part A - Pharmacokinetic of KAE609: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Tmax was calculated from plasma concentration-time data using non-compartmental methods based on the actual time of sample collection and summarized using descriptive statistics.
Time Frame: Day 1 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hour (hr) | 0.167 [0.0167 to 0.167] | 0.0333 [0.0333 to 0.217] | 0.333 [0.183 to 0.550] | 0.167 [0.167 to 0.183] | 0.167 [0.167 to 0.200]

4. Secondary Outcome: Part A - Pharmacokinetic of KAE609: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. AUClast was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Day 1 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 2690 (977) | 9540 (1640) | 25400 (1770) | 53700 (20900) | 60800 (11600)

5. Secondary Outcome: Part A - Pharmacokinetic of KAE609: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. AUCinf was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Day 1 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 2770 (990) | 9750 (1730) | 25600 (1730) | 57400 (22100) | 62000 (11500)

6. Secondary Outcome: Part A - Pharmacokinetic of KAE609: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC0-24hrs)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. AUC0-24hrs was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Day 1 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 1450 (330) | 4540 (673) | 13500 (2230) | 23200 (7920) | 26200 (3600)

7. Secondary Outcome: Part A - Pharmacokinetic of KAE609: Terminal Elimination Half-life (T1/2)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. T1/2 was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Day 1 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour (hr)
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hour (hr) | 27.7 (8.89) | 30.5 (6.79) | 21.9 (6.76) | 38.9 (12.8) | 29.4 (5.39)

8. Secondary Outcome: Part A - Pharmacokinetic of KAE609: Clearance From Plasma (CL) Following Drug Administration
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. CL was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Day 1 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter/hour (mL/h)
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Milliliter/hour (mL/h) | 4330 (1890) | 3150 (507) | 2940 (192) | 2430 (1120) | 3500 (700)

9. Secondary Outcome: Part A - Pharmacokinetic of KAE609: Apparent Volume of Distribution During Terminal Phase (Vz)
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Vz was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Day 1 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Milliliter (mL) | 154000 (20400) | 138000 (34000) | 92900 (29600) | 124000 (32700) | 151000 (50400)

10. Secondary Outcome: Part B - Pharmacokinetic of KAE609: Maximum Observed Plasma Concentration (Cmax)
Description: as for outcome 2
Time Frame: Days 1 and 5 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg)
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 1 | 3920 (999) | 4530 (705)
  Day 5 | 4630 (2670) | 5540 (2090)

11. Secondary Outcome: Part B - Pharmacokinetic of KAE609: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: as for outcome 3
Time Frame: Days 1 and 5 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg)
Number analyzed (Participants) | 6 | 6
Hour (hr)
  Day 1 | 0.100 [0.0333 to 0.500] | 0.167 [0.167 to 0.183]
  Day 5 | 0.0333 [0.0333 to 0.167] | 0.167 [0.167 to 0.167]

12. Secondary Outcome: Part B - Pharmacokinetic of KAE609: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Description: as for outcome 4
Time Frame: Day 5 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg)
Number analyzed (Participants) | 6 | 6
h*ng/mL | 58500 (23000) | 121000 (56100)

13. Secondary Outcome: Part B - Pharmacokinetic of KAE609: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC0-24hrs)
Description: as for outcome 6
Time Frame: Days 1 and 5 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg)
Number analyzed (Participants) | 6 | 6
h*ng/mL
  Day 1 | 13200 (1770) | 16500 (2290)
  Day 5 | 20000 (4890) | 40600 (11400)

14. Secondary Outcome: Part B - Pharmacokinetic of KAE609: Terminal Elimination Half-life (T1/2)
Description: as for outcome 7
Time Frame: Days 1 and 5 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour (hr)
Arm/Group | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg)
Number analyzed (Participants) | 6 | 6
Hour (hr)
  Day 1 | 25.0 (8.16) | 18.1 (2.83)
  Day 5 | 35.5 (8.58) | 31.9 (12.5)

15. Secondary Outcome: Part B - Pharmacokinetic of KAE609: Clearance From Plasma (CL) Following Drug Administration
Description: as for outcome 8
Time Frame: Day 5 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter/hour (mL/h)
Arm/Group | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg)
Number analyzed (Participants) | 6 | 6
Milliliter/hour (mL/h) | 3140 (717) | 3160 (907)

16. Secondary Outcome: Part B - Pharmacokinetic of KAE609: Apparent Volume of Distribution During Terminal Phase (Vz)
Description: as for outcome 9
Time Frame: Day 5 (-1 hr, 2 min, 10 min, 30 min, 1 hr, 3 hr, 6 hr, 12 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg)
Number analyzed (Participants) | 6 | 6
Milliliter (mL) | 175000 (14700) | 173000 (29700)

ADVERSE EVENTS:
Time Frame: On-treatment Adverse events (AEs) and serious AEs (including the All-Cause Mortality data table) are presented from first dose of study treatment until last dose of study treatment plus 30 days post treatment, assessed for up to 4 months.
Description: Any sign or symptom that occurs during the treatment period plus 30 days post-treatment.
Arm/Group | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg) | Part A (Single-ascending Dose (SAD): Pooled KAE609 | Part A (Single-ascending Dose (SAD): Pooled Placebo | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg) | Part B (Multiple-ascending Dose (MAD): Pooled KAE609 | Part B (Multiple-ascending Dose (MAD): Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/30 | 0/9 | 0/6 | 0/6 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 1/30 | 0/9 | 0/6 | 0/6 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 1/6 | 2/6 | 6/6 | 10/30 | 5/9 | 4/6 | 6/6 | 10/12 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) (N=6) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) (N=6) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) (N=6) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) (N=6) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg) (N=6) | Part A (Single-ascending Dose (SAD): Pooled KAE609 (N=30) | Part A (Single-ascending Dose (SAD): Pooled Placebo (N=9) | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) (N=6) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg) (N=6) | Part B (Multiple-ascending Dose (MAD): Pooled KAE609 (N=12) | Part B (Multiple-ascending Dose (MAD): Pooled Placebo (N=6)
Testicular embryonal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular malignant teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Single-ascending Dose (SAD): Cohort A1 (KAE609 10.5 mg) (N=6) | Part A (Single-ascending Dose (SAD): Cohort A2 (KAE609 30 mg) (N=6) | Part A (Single-ascending Dose (SAD): Cohort A3 (KAE609 75 mg) (N=6) | Part A (Single-ascending Dose (SAD): Cohort A4 (KAE609 120 mg) (N=6) | Part A (Single-ascending Dose (SAD): Cohort A5 (KAE609 210 mg) (N=6) | Part A (Single-ascending Dose (SAD): Pooled KAE609 (N=30) | Part A (Single-ascending Dose (SAD): Pooled Placebo (N=9) | Part B (Multiple-ascending Dose (MAD): Cohort B1 (KAE609 60 mg) (N=6) | Part B (Multiple-ascending Dose (MAD): Cohort B2 (KAE609 120 mg) (N=6) | Part B (Multiple-ascending Dose (MAD): Pooled KAE609 (N=12) | Part B (Multiple-ascending Dose (MAD): Pooled Placebo (N=6)
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Catheter site oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Infusion site discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 3 | 4 | 7 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 4 | 3 | 2 | 3 | 5 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Semen discolouration (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT04321252/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT04321252/SAP_001.pdf